CLINICAL TRIAL: NCT00885027
Title: Quality of Life in Patients With BPH and Nocturia Before and After Tamsulosin Ocas® Treatment
Brief Title: MEN STUDY (ESTUDIO MEN) Quality of Life in Patients With BPH and Nocturia Before and After Tamsulosin Ocas® Treatment
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 527.80
Record Dates: First submitted 2009-01-20; First posted 2009-04-21 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This is an exploratory study, to evaluate the improvement in terms of quality of life that can be reached by a group of outpatients with BPH ( Benign Prostatic Hyperplasia ) and nocturia when they are under treatment with Secotex Ocas.

This study will explore, the progress in terms of quality of life that can be reached by a group of outpatients with BPH ( Benign Prostatic Hyperplasia) and nocturia treated with Secotex OCAS®.

This is a not controlled study, " before and after type", which will consist of an assessment, of the quality of life for outpatients with BPH symptoms including nocturia, through the use of the Spanish version of the Nocturia Quality-of-life (NQoL) questionnaire, at three different moments:

1. Before to start Secotex OCAS® treatment.
2. Thirty (30) days after first visit and starting Secotex OCAS® treatment
3. Ninethy (90) days after first visit and starting Secotex Ocas® treatment

DETAILED DESCRIPTION:
Study Design:

ELIGIBILITY:
Inclusion Criteria:

Men 40 years old with benign prostatic hyperplasia (BPH) which, according their doctor, requires medical treatment to improve quality of life. Patients may be new in the treatment or can be treated with other medicines but not having responded adequately to treatment (Not should be taking Tamsulosin OCAS).

PSA < 4.0 ng/ml or 4 ¿ 10ng/ml with prior negative Transrectal biopsy. IPSS > 12 points. Two or more episodes of nocturia per night (score equal or exceed 2 in question 7 of IPSS).

IPSS QoL (Question 8) > 3 points (score equal or superior to 3 in question 8 of Quality of Life (QoL) of IPSS).

Acceptance written of their participation in the study by the informed consent. The decision of treatment should be based on the best clinical practice accepted standard and according to the information for prescription for Secotex OCAS® 0.4 mg.

Exclusion Criteria:

Patients with clear indication to receive surgical treatment Hospitalized patients Patients with physical or mental disabilities that prevent, even with the help of doctor, completing the instruments of assessment of the survey Patients with a history of malignant disease Patients with known hypersensitivity to tamsulosin or to another component of the product Patients with a history of orthostatic hypotension or severe liver failure Positive digital rectal test for possible neoplasia or biochemical evidence of high PSA with figures > 4.0 ng/ml Patients with diastolic blood pressure less than 60 mmHg or tachycardia greater to 120 beats per minute

Other reasons for the exclusion:

* Acute Urinary Retention (AUR)
* Urinary tract infection
* Renal failure

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: men >=40 years old with BPH
Sampling Method: Probability Sample
Enrollment: 1342 (Actual)
Dates: Start 2009-03; Primary Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Reductions in the intensity of symptoms, evaluated using the IPSS scale. | up to 90 days
Improvement in quality of life, measured using the NQoL questionnaire. | up to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (18):
- Colombia (18):
  - Boehringer Ingelheim Investigational Site, Barranquilla
  - Boehringer Ingelheim Investigational Site, Bogotá
  - Boehringer Ingelheim Investigational Site, Boyacá
  - Boehringer Ingelheim Investigational Site, Bucaramanga
  - Boehringer Ingelheim Investigational Site, Cali
  - Boehringer Ingelheim Investigational Site, Cartagena
  - Boehringer Ingelheim Investigational Site, Cúcuta
  - Boehringer Ingelheim Investigational Site, Ibagué
  - Boehringer Ingelheim Investigational Site, Manizales
  - Boehringer Ingelheim Investigational Site, Medellín
  - Boehringer Ingelheim Investigational Site, Palmira
  - Boehringer Ingelheim Investigational Site, Pereira
  - Boehringer Ingelheim Investigational Site, Popayán
  - Boehringer Ingelheim Investigational Site, Santa Marta
  - Boehringer Ingelheim Investigational Site, Sincelejo
  - Boehringer Ingelheim Investigational Site, Tuluá
  - Boehringer Ingelheim Investigational Site, Valledupar
  - Boehringer Ingelheim Investigational Site, Villavicencio